CLINICAL TRIAL: NCT01372124
Title: A Phase I, Open Label, Parallel Group, Multi-center Single Dose Trial to Evaluate the Effect of Renal Impairment on Pharmacokinetics of NOX-E36
Brief Title: A Phase I Clinical Trial to Evaluate the Effect of Renal Impairment on Pharmacokinetics of NOX-E36
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TME Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNOXE36C201
Record Dates: First submitted 2011-06-08; First posted 2011-06-13 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Renal Impairment
Keywords: Renal impairment; NOX-E36
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NOX-E36 (Experimental): All subjects included in this study will receive the same dose of NOX E36.
  Interventions: Drug: NOX-E36

INTERVENTIONS:
Drug: NOX-E36 — All subjects included in this study will receive the same dose of NOX E36. In previous clinical trials, single intravenous doses of NOX E36 up to 2 mg/kg body weight and single subcutaneous doses of up to 0.5 mg/kg body weight appeared to be safe and well tolerated in healthy volunteers. Pharmacokinetic analyses have shown dose linearity

SUMMARY:
This is a multi center, open label, parallel group, single administration, phase I trial, in subjects with mild, moderate or severe renal impairment and a control group with normal renal function.

DETAILED DESCRIPTION:
Current diabetes therapy does not stop progression of the disease and the development of diabetes mellitus (DM)-associated complications. A major concern in DM-patients is renal impairment due to nephropathy leading to a reduced glomerular filtration rate (GFR). It has been established that chronic (sub)clinical inflammation is crucial for the onset and progression of DM.

CCL2, also known as Monocyte chemoattractant protein 1 (MCP 1) is a chemokine from the cysteine-cysteine family, secreted by leukocytes or tissue cells. CCL2 promotes monocyte emigration from the bone marrow, activates monocytes and macrophages and directs their migration to sites of inflammation. Recent animal studies and clinical trials indicate a critical involvement of CCL2 in DM and diabetic nephropathy, suggesting that CCL2 may be a potential target for therapeutic intervention in DM. Finally, protein overload and oxidative challenge of the diseased kidney was suggested to stimulate CCL2 expression in renal tubuli, thereby accelerating the progression of diabetic nephropathy.

As NOX E36 is designed to specifically target human MCP-1/CCL2. This study is performed to evaluate the role of renal impairment for adequate dosing recommendations in the planned target population.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects (age 18-75 years, both inclusive)
2. Male subjects who agree to sexual abstinence and/or use a highly effective method of birth control. Female partners of male subjects must be of non-child bearing potential or must practice an adequate non-hormonal contraceptive method to prevent pregnancies.
3. Subjects will be categorized as follows based on creatinine clearance(mL/min/1.73m2): Normal renal function: CrCl > 80; mild renal impairment: 50 ≤ CrCl ≤ 80; moderate renal impairment: 30 ≤ CrCl ≤ 50; severe renal impairment: CrCl < 30
4. Body Mass Index (BMI) between 22 and 40 kg/m², both inclusive.

Exclusion Criteria:

1. Women of childbearing potential
2. Patients who have received kidney transplantation.
3. Patients receiving hemodialysis to control their disease.
4. Any clinically significant abnormality other than related to the renal impairment following the investigator's review of the physical examination, ECG and clinical laboratory tests at screening.
5. Not able to communicate meaningfully with the investigator and staff.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Boris Sazu, MD, Principal Investigator — INNOPHAR MO s.R.L.; Éva Péterfai, Principal Investigator — DRC
Locations (2):
- DRC, Balatonfüred, Hungary
- Innophar Mo S.R.L., Chisinau, Moldova